CLINICAL TRIAL: NCT02054910
Title: Randomized Single Blinded Control Trial Comparing EUS Guided Celiac Plexus Block (CPB) Versus Sham Treatment for Pain Management in Small Duct Chronic Pancreatitis
Brief Title: CPB Versus Sham Treatment for Pain Management in Small Duct Chronic Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Charles Mel Wilcox, MD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F130822012
Record Dates: First submitted 2014-01-29; First posted 2014-02-04 (Estimated); Results first posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Celiac Plexus Block (Experimental): Celiac Plexus Block will be administered following EUS
  Interventions: Procedure: Celiac Plexus Block
- Sham (Sham Comparator): A celiac plexus block will not be administered for pain management
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: Celiac Plexus Block — Patients will receive celiac plexus block during endoscopy.
  Arms: Celiac Plexus Block
Procedure: Sham — Patients will not receive celiac plexus block during endoscopy.
  Arms: Sham

SUMMARY:
This study assesses the pain response to Endoscopic Ultrasound (EUS) guided Celiac Plexus Block (CPB) treatment in comparison to EUS without a pain block administered. All participants will receive medications for pain as needed.

DETAILED DESCRIPTION:
The purpose of this study is to assess pain response to EUS guided celiac plexus block treatment compared to no treatment. The Visual Analog Scale (VAS) is the primary measure. Secondary aims include the comparison of quality of life scores, need for narcotics, to assess the effect of EUS-CPB on overall mental state using the Beck's Depression Index, and to assess the effect of EUS-CBP on health care utilization and on employment.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred to UAB Endoscopy Unit for with known chronic pancreatitis
* Patients referred to the endoscopy unit with abdominal pain with suspicion of chronic pancreatitis meeting 5 of 9 parenchymal and ductal changes (i.e. lobulations, hyperechoic stranding, hyperechoic foci, cysts, calcification, irregular duct, hyperechoic walls, side branch dilations and ductal calculi).

Exclusion Criteria:

* Age <19 years
* Unable to safely undergo EUS for any reason
* Coagulopathy (INR >1.6, Prothrombin Time >18secs, Thrombocytopenia <80,000 cells/ml)
* Unable to consent
* Non-English speaking patients.
* Previously undergone CPB
* Pregnancy and Breast feeding
* Patients with ductal strictures, calcification, pancreatic ductal calculi, pseudocysts.
* Previous pancreatic surgery
* Previous pseudocyst drainage
* Other documented causes of abdominal pain.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Wilcox, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Celiac Plexus Block: Celiac Plexus Block will be administered following EUS
  Celiac Plexus Block
- Sham: A celiac plexus block will not be administered for pain management
  Sham
Period: Overall Study
Arm/Group | Celiac Plexus Block | Sham
Started | 4 | 1
Completed | 0 | 0
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celiac Plexus Block | Sham | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 1 | 1 | 2
Gender [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Response Over a 6 Month Period of Time Using the VAS Score
Description: Pain scores will be assessed by comparing the mean number change using the Visual Analog Scale (VAS) from baseline to 6 month. The scale is 10 - 0, with 10 being agonizing pain and 0 being no pain.
Time Frame: baseline to 6 months
Population: All subjects were lost to follow up by 6 months; the primary endpoint was not collected for any subject
Arm/Group | Celiac Plexus Block | Sham
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Mean Quality of Life Score Between Each Group at 6 Months
Description: The American Chronic Pain Association, Quality of Life Score will be used. This scoring ranges from 0 (Stay in bed all day Feel hopeless and helpless about life - non-functioning) to 10 (Go to work/volunteer each day Normal daily activities each day Have a social life outside of work Take an active part in family life - normal life).
Time Frame: 6 months post baseline
Population: All subjects were lost to follow up by 6 months; the secondary endpoint was not collected for any subject
Arm/Group | Celiac Plexus Block | Sham
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Subject in Each Group Requiring Administration of Narcotics During 6 Months Post Baseline
Description: the number of subjects receiving a narcotic drug during the 6 months post baseline will be noted.
Time Frame: baseline to 6 months
Population: All subjects were lost to follow up by 6 months; the secondary endpoint was not collected for any subject
Arm/Group | Celiac Plexus Block | Sham
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mean Mental State Between Groups Using the Beck's Depression Index at 6 Months.
Description: The Beck's Depression scale was used to indicate subject's depression:
  0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression.
Time Frame: baseline to 6 months
Population: All subjects were lost to follow up by 6 months; the secondary endpoint was not collected for any subject
Arm/Group | Celiac Plexus Block | Sham
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Mean Number of Times Subjects in Each Group Accessed the Health Care System Within 6 Months Post Procedure
Description: The number of times each subject accessed the health care system will be collected, and then the mean will be calculated for each group
Time Frame: baseline to 6 months
Population: All subjects were lost to follow up by 6 months; since everyone dropped out at different times before the 6 month point, the data would not be evaluable.
Arm/Group | Celiac Plexus Block | Sham
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: % of Subjects in Each Group That Are Employed at 6 Months Post Procedure.
Description: Subjects will be asked about employment at 6 months post procedure
Time Frame: baseline to 6 months
Population: All subjects were lost to follow up by 6 months; the secondary endpoint was not collected for any subject
Arm/Group | Celiac Plexus Block | Sham
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24-48 hour, 2 week, 6 month, 12 month
Arm/Group | Celiac Plexus Block | Sham
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 0/4 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes